CLINICAL TRIAL: NCT04479657
Title: A Randomized Controlled Study of Qingfei Granule for the Treatment of the Pediatric Acute Upper Respiratory Tract Infection With Bacterial Infection
Brief Title: Qingfei Granule for the Treatment of the Pediatric Acute Upper Respiratory Tract Infection With Bacterial Infection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhong Wang (Other)
Responsible Party: Sponsor-Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QFKL V3.0
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Upper Respiratory Tract Infection; Bacterial Infection; Chinese Medicine; Pediatric Acute Upper Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections; Bacterial Infections | interventions — Cefuroxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QingFei Granule+Cefuroxime group (Experimental): Cefuroxime：30mg/kg/d,bid QingFei Granule: tid
  Interventions: Drug: QingFei Granule; Drug: Cefuroxime
- Cefuroxime group (Active Comparator): Cefuroxime：30mg/kg/d,bid
  Interventions: Drug: Cefuroxime

INTERVENTIONS:
Drug: QingFei Granule — QingFei Granule is made from 6 commonly herbal medicine granule, such as Jingjie,Huang Qin,Lianqiao,etc. The children were given one package of QingFei Granule every day, dividing into 3 times to be administrated. It's be given for 5 days.
  Arms: QingFei Granule+Cefuroxime group
Drug: Cefuroxime — 30mg/kg/d,bid, used until to the normalization of blood routine。

SUMMARY:
The study aims to assess the antibacterial effect and symptoms-relief of Qingfei Granule in the patients with pediatric acute upper respiratory tract infection with bacterial infection.

DETAILED DESCRIPTION:
Upper respiratory tract infection is the most common respiratory disease in childhood, and the incidence rate accounts for more than 60% of pediatric outpatients, ranking first in pediatric diseases. At present, antibiotics are commonly used to treat children with upper respiratory tract infections. However, due to the large amount of clinical use of antibiotics in recent years, the resistance of various pathogens has become stronger and stronger, which has caused the majority of clinicians and researchers to turn their attention to traditional Chinese medicine. Qingfei Granule is composed of six common herbal medicines such as Schizonepeta (Jing-Jie),Radix Scutellariae (Huang-qin),Forsythia (Lian-Qiao), etc. After upper respiratory tract infections with bacterial infections, chills, fever, runny nose, red and sore throat may occur, and may be accompanied by mild cough, thin red tongue, yellow moss, floating pulse,which is considered as the exogenous wind-heat Zheng in Chinese medicine. The study aims to assess the antibacterial effect and symptoms-relief of Qingfei Granule in the patients with pediatric acute upper respiratory tract infection with bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis with the acute upper respiratory tract infection;
2. Diagnosis with wind-heat Zheng according to Chinese medicine;
3. Age: 5-14 years old;
4. Body temperature ≥ 37.5 ℃;
5. White blood cell count> 12 × 10^9 / L, and / or neutrophil ratio over than 70%;
6. The informed consent process complies with the regulations, and the legal agent or the child (≥8 years old) jointly sign the informed consent

Exclusion Criteria:

(1) Acute bacterial otitis media; (2) Patients with periodontitis or periodontal abscess (3) Candidiasis; (4) Patients with positive mycoplasma; (5) Taking antibiotics, anti-inflammatory drugs, and antihistamines; (6) Patients with severe comorbidities of heart, liver and kidney; (7) Other patients with acute infectious diseases and mycoplasma pneumoniae infections with symptoms similar to upper respiratory tract infection; (8) Children with a history of epilepsy or convulsions; (9) Patients with mental illness; (10) Those who are allergic to treatment drugs; (11) Participated in other clinical trials in the past month; (12) The investigator evaluates that it is not suitable to participate in this clinical trial or according to the investigator's judgment, who is likely to loss to follow-up.

-

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-10-17 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Bacterial clearance | 0, Day 5
  The pharyngeal swabs were used for sampling, and the pharyngeal flora diversity amplicon sequencing was used to analyze the pharyngeal flora spectrum, and the change of pathogenic bacteria flora spectrum before and after treatment was analyzed to qualitatively judge the bacterial clearance.
  Calculate the bacterial clearance rate = (number of people removed / total number of people tested) × 100%

SECONDARY OUTCOMES:
Clinical remission rate of disease | Day 3,Day 5
  The clinical remission rate of disease is defined as: the main symptoms such as chills, fever, nasal congestion, runny nose, sore throat, cough, etc. alleviate or disappear. Upper respiratory tract infection symptom scale score decreased by more than 70% compared with baseline
Fever clearance time | Up to Day 5
  record once every 4 to 8 h after treatment.
Treatment failure rate | Up to Day 5
  Treatment failure is defined as: body temperature does not decrease for 3 consecutive days, and / or complicated by laryngitis, tracheobronchitis, pneumonia, myocarditis, and / or oral antibiotics are switched to intravenous antibiotics.
The incidence of the complications | Up to Day 5
  complicated with laryngitis, tracheo-bronchitis, pneumonia, myocarditis and other complications
The usage of the ibuprofen | Up to Day 5
  If the temperature is over 38.5℃ or the child feel unbearable discomfort, the child will be given with ibuprofen. The usage of the ibuprofen (including the usage times and detail amount will be recorded in the patients' dairy.
The usage of antibiotics (Cefuroxime) | Up to Day 5
  The usage of Cefuroxime (including the usage times and detail amount will be recorded in the patients' dairy.
The normalization rate of the blood routine | Day 3, Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Dongfang Hospital, Beijing, Beijing Municipality, China